CLINICAL TRIAL: NCT06734936
Title: The Effect of Video Viewing With Virtual Reality Glasses on Pain and Anxiety During Urethral Bladder Catheterization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Selcuk Ozturk, Principal İnvestigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ErciyesU bladdercathetersgg38
Record Dates: First submitted 2023-12-27; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): SGG applied group
  Interventions: Other: Playing videos with sgg
- control group (No Intervention): sgg unused group

INTERVENTIONS:
Other: Playing videos with sgg — Playing videos with sgg
  Arms: experimental group

SUMMARY:
Urinary catheterization is an interventional practice performed by placing a urinary catheter, which is a latex, polyurethane or silicone tube, into the bladder through the patient's urethra to evacuate the urine accumulated in the bladder for diagnosis and treatment purposes. Urinary catheterization is one of the most frequently used procedures in emergency departments. A urinary catheter is applied at least once to 5-11% of patients applying to the emergency department. Urinary catheter in emergency departments; It is applied for acute or chronic urinary retention, relief of urinary tract obstruction, determination of residual urine amount, prostate hyperplasia, drainage of hypotonic bladder, neurogenic bladder, urdodynamic examinations, contrast radiological examination, obtaining sterile urine sample and bladder irrigation in hematuria. Pain and anxiety are among the common symptoms in patients undergoing urinary catheterization.

During the urinary catheterization procedure, 2% lidocaine gel is the most commonly used agent and is applied in an average amount of 6-10 ml. Since the procedure area is still sensitive despite appropriate local anesthesia, patients cannot be completely prevented from experiencing pain and anxiety . When the literature is scanned, it is reported that 75.4-95.3% of patients who underwent urinary catheterization experience pain, and that this pain is at moderate to severe levels in approximately 41.2-88.7% of the patients . Yücel found the frequency of anxiety in patients who underwent urinary catheterization to be 85%, and it was determined that 37% of this anxiety was mild, 64% was moderate, and 79% was severe .

In addition to local anesthesia, parecetemol and dexketoprofen derivative painkillers can be administered orally, intramuscularly and intravenously to control pain and anxiety that may develop during and after the urinary catheterization procedure. It has been shown that these pharmacological methods used in pain and anxiety control reduce pain and anxiety in patients, but may cause some side effects such as hypotension, bradycardia, nausea and vomiting, skin rash, itching, increase the need for auxiliary personnel and equipment, and prolong the patient's hospital stay.

Nurses who are with the patient for a long time have a major role in reducing pain and anxiety. In painful interventional procedures such as urinary catheterization, some non-pharmacological methods are applied by nurses to prevent pain and anxiety. In this context, practices such as music therapy and hypnosis are used . Apart from music and hypnosis, another non-pharmacological method that can be used to control pain and anxiety is Virtual Reality Glasses (VR). VR, one of the methods of diverting attention, is an advanced form of human-computer interaction that allows people to hear the sounds and stimuli accompanying the visual landscape through headphones, allowing the person to feel in another world by moving away from the hospital . Research conducted with SGG shows that virtual reality is an effective method for pain control , post-burn physiotherapy, outpatient chemotherapy treatment , port insertion, lumbar puncture, labor pain , AVF cannulation and breast biopsy , the video watched with SGG has been shown to reduce pain and anxiety. It has been shown to be effective on There is no study in the literature showing the effect of SGG use on pain and anxiety control during urinary catheter procedure.

The aim of our study is to reveal the effect of virtual reality glasses on pain and anxiety in patients undergoing urinary catheter procedure. A limited amount of literature reports that virtual reality glasses are effective in controlling pain and anxiety before and during various interventional procedures. In this context, as researchers, the investigators believe that this is a study with high original value.

DETAILED DESCRIPTION:
GENERAL INFORMATION Urinary Catheterization Urinary catheterization is the process of inserting a catheter from the urinary tract into the bladder . Urinary catheterization is frequently used both in and outside the hospital. Approximately one quarter of hospitalized individuals undergo urinary catheterization . Although 15-25% of hospitalized patients have a urinary catheter applied at least once, this rate increases to 75-90% in intensive care patients . However, it has been observed that urinary catheter insertion rates have increased recently.

Catheter Selection in Urinary Catheterization Since the catheter may cause trauma due to the effect of a foreign body, a small diameter catheter suitable for the patient and the purpose of the application should be selected. A catheter size of 12-14 Fr should be used in women and 14-16 Fr in men . If the urine is very cloudy and concentrated, a larger diameter catheter can be selected to ensure easier drainage. The catheter balloon is inflated by administering the amount of sterile fluid written on the selected catheter.

Indications for Urinary Catheterization Urinary catheterization should be performed in the presence of the following indications, and the urinary catheterization process should be terminated when the presence of the indication is eliminated by constant questioning.

* Acute urinary retention,
* Urinary obstructions,
* Surgical procedure on organs adjacent to the genito-urinary system,
* Prolongation of the duration of the surgical procedure
* Individuals who receive high-dose infusion or receive diuretic medication during the surgical procedure,
* Critical situations where urine output must be calculated hourly,
* Situations where urine output needs to be monitored during the surgical procedure,
* Individuals with incontinence problems who have open perineal or sacral pressure sores,
* Individuals who need to remain immobile for a while,
* Intravesical treatment,
* Accumulating urine in the bladder for diagnostic purposes Complications Associated with Urinary Catheterization Urinary catheterization is a procedure that causes many complications in hospitalized patients. Some complications and their causes due to urinary catheterization are explained below.

  * Pain
  * Trauma
  * Scaling
  * Hematuria
  * Bladder spasm
  * incontinence
  * Urinary System Infection Nursing Care in Urinary Catheterization Urinary catheterization is a procedure performed under the responsibility of a nurse upon the request of a doctor, and its application and removal is a complicated nursing practice. It is very important for the catheterization procedure to be carried out in accordance with surgical aseptic technique to protect the sterile urinary system. Many complications may develop after a urinary catheter is not installed under appropriate conditions and the health status of the individual may be negatively affected . The most common complication seen during urinary catheterization is CI-UTI. Complications seen after the catheterization process is terminated are UI and urinary retention . In practice, it is necessary to evaluate the individual's needs with a humanistic and holistic approach, determine the indication, and perform nursing care with the correct technique .

Studies Examining the Role of Sgg in Pain and Anxiety Control Schneider showed 16 breast cancer patients aged 50 and over watching submarine, titanic and museum tour videos with SGG during chemotherapy treatment and found that there was a significant decrease in fatigue, anxiety and perception of time passed during chemotherapy. In another study, it was reported that the pain felt during the dressing process decreased in 36 burn patients using SGG . Gershon determined that CSR was an effective distraction technique in reducing pain and reduced anxiety during interventional procedures in cancer patients between the ages of 7-19. Espinoza showed 33 cancer patients between the ages of 41 and 85 who were undergoing chemotherapy treatment, watching nature and park videos for 30 minutes with SGG, and determined that after the application, the patients' anxiety levels decreased and their happiness levels increased. In their study, Jahani Shoorab examined the effect of SGG on pain during episiotomy repair with 30 primiparous patients; They determined that there was a statistically significant difference between the pain score during episiotomy repair in both groups and that SGG was an effective complementary non-pharmacological method to reduce pain during episiotomy repair. In their study, Glenon examined the effect of SGG on pain and anxiety in patients undergoing CIAB; It revealed that there was no statistically significant decrease in pain and anxiety in the SGG group. However, it was reported that there was a similar decrease in pain and anxiety levels in the experimental and control groups before and after the procedure.

In their study where Veldhuijzen evaluated the effect of SGG to relieve pain and discomfort during colonoscopy, they found that patient comfort, pain, anxiety and satisfaction regarding the procedure were similar in the group using and not using SGG.

In their study, De Araújo examined the effect of SGG application on pain during chronic wound dressing change; It has been shown that SGG has positive effects in relieving pain and there is a decrease in pain scores before and after dressing.

Burn debridement , chemotherapy applications , peripheral intravenous catheterization , lumbar puncture , dental treatment Studies have reported that SGG use has positive effects on pain and anxiety scores.

MATERIALS AND METHODS 3.1. Purpose and Form of the Research This research was planned as a randomized controlled experimental study to reveal the effect of video viewing with virtual reality glasses on pain and anxiety during urethral bladder catheterization. Stratified randomization in terms of age and gender will be applied using a computer program to determine patient groups. The reason for applying stratified randomization in terms of age and gender is to ensure equal distribution of age and gender factors that may affect the study results across groups.

Population and Sample of the Research The accessible sample of the study will consist of patients between the ages of 18 and 65 who applied to Kayseri City Training and Research Hospital Emergency Service and requested bladder catheterization. The population of the randomized controlled study will be determined by excluding individuals from the accessible sample according to the exclusion criteria of the study. In determining the number of samples, a comparison of two groups, SGG and control, will be made using the G.Power 3.1 package program. For the sample size of the study, taking into account the results of similar studies, it was planned to recruit a total of 80 patients, 40 in the control group and 40 in the virtual reality glasses (VRG) group. Randomized controlled study groups will be created by random selection from the calculated individuals using a simple random numbers table with the help of the Excel program. It was planned to select intervention groups and control groups by random assignment to individuals in the randomized controlled study groups.

Criteria for Inclusion in the Study The scope of the research; Those between the ages of 18 and 65, Clinically stable and easy to communicate with, Able to communicate in Turkish, Having no psychiatric, mental, visual or hearing problems, Does not have any discomfort that would prevent him from lying in the supine position, Individuals who agree to participate in the research will be included.

Exclusion Criteria in the Study The scope of the research; For women who have given birth twice or more, Having a history of gynecological surgery, Having a history of prostate cancer, Those with prostate hyperplasia Having a history of urological surgery, More than 2 attempts to apply a urinary catheter, Those who have pain before the procedure and use any analgesic medication, Using anxiolytic and/or sedative drugs, Individuals who do not agree to participate in the research will not be included.

Termination Criteria for the Study Clinically unstable during the procedure, Patients who want to remove the catheter due to anxiety or pain during the procedure, They will be identified as patients who wish to withdraw from the study.

Research Variables Dependent Variables: Scores from VAS and State-Trait Anxiety Scale, vital signs constitute the dependent variables of the study.

Independent Variables: Descriptive characteristics of the individuals participating in the research (such as age, gender) and the application of watching videos with virtual reality glasses constitute the independent variables of the research.

Data Collection Forms and Tools In collecting research data, the Patient Introduction Form , Informed Voluntary Consent Form was created by the researcher to determine the patient's descriptive and medical characteristics by scanning the relevant literature, and Visual Analogue Scale (VAS) was used to evaluate the severity of pain , State and Trait Anxiety Scale , SGG were used to determine the anxiety level.

Patient Introduction Form: The patient introduction form, prepared by the researcher by reviewing the relevant literature, includes data about the patients' socio-demographic characteristics such as age, gender, education level, profession, marital status, income status, and disease-related characteristics . The Patient Introduction Form will be filled out by meeting the patients face to face and using the patient file.

Informed Volunteer Consent Form: "Informed Volunteer Consent Form" will be used to inform all individuals participating in the research about the research and to indicate that they accept their participation in the research.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18 and 65,
* Clinically stable and easy to communicate with,
* Able to communicate in Turkish,
* Having no psychiatric, mental, visual or hearing problems,
* Does not have any discomfort that would prevent him from lying in the supine position,
* Individuals who agree to participate in the research will be included.

Exclusion Criteria:

* For women who have given birth twice or more,
* Having a history of gynecological surgery,
* Having a history of prostate cancer,
* Those with prostate hyperplasia
* Having a history of urological surgery,
* More than 2 attempts to apply a urinary catheter,
* Those who have pain before the procedure and use any analgesic medication,
* Using anxiolytic and/or sedative drugs,
* Individuals who do not agree to participate in the research will not be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
STATE AND TRAITING ANXIETY SCALE | UP TO 8 WEEKS
  STATE AND TRAIT ANXIETY SCALE SCORING Manual Scoring: Two separate keys are prepared for each of the direct and reverse statements. Thus, the total weights of the direct statements are calculated with one key and the total weights of the reversed statements are calculated with the second key. The total weighted score for the direct statements is subtracted from the total weighted score for the reversed statements.
  A predetermined and unchanging value is added to this number. This constant value is 50 for the State Anxiety Scale and 35 for the Trait Anxiety Scale. The value obtained is the anxiety score of the individual.

SECONDARY OUTCOMES:
VISUAL ANALOGUE SCALE (VAS) | UP TO 8 WEEKS
  Determines the score between '0' No Pain - '10' Most excruciating pain scale Visual Analog Scale (VAS) cannot be measured numerically is used to convert some values into numerical form. At the two ends of a 100 mm line The two extreme definitions of the parameter to be evaluated are written and the patient is asked to draw his/her own line on this line.
  by drawing a line or putting a dot or marking where the situation is appropriate to indicate the pain. For example, for pain, at one end, I have no pain, and at the other end, I have very severe pain.
  The pain is written and the patient marks his/her current state on this line. No pain at all the length of the distance from the place where the patient is absent to the place marked by the patient indicates pain.

IPD SHARING:
Plan to Share IPD: Undecided